CLINICAL TRIAL: NCT01696370
Title: A Phase 2b Randomised, Double Blind, Placebo-controlled Trial of Trimetazidine Therapy in Patients With Non-obstructive Hypertrophic Cardiomyopathy
Brief Title: Trimetazidine Therapy in Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/0216
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2011-08

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Trimetazidine
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trimetazidine (Active Comparator)
  Interventions: Drug: Trimetazidine
- Placebo capsule (Placebo Comparator)
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Drug: Trimetazidine — Trimetazidine 20mg three times per day for 3 months
  Arms: Trimetazidine
Other: Placebo capsule — one capsule three times per day for 3 months
  Arms: Placebo capsule

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a common inherited heart condition that causes breathlessness, chest pain and fatigue. There are few treatments available. The investigators have recently shown that a drug called perhexiline reduced symptoms and improved exercise capacity in patients with HCM. This change appears to be driven by alterations in myocardial energy metabolism. The aim of this trial is to test a similar drug, trimetazidine, in a group of symptomatic patients with non-obstructive HCM.

HYPOTHESIS: trimetazidine will improve symptoms, peak oxygen consumption, cardiac function and arrhythmia burden in medically refractory symptomatic patients with non-obstructive HCM.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertrophic cardiomyopathy (HCM) is a common inherited disorder of heart muscle affecting 1 in 500 individuals worldwide. It is associated with arrhythmias, heart failure and sudden death in young people. In the majority of patients, HCM is caused by mutations in genes encoding cardiac contractile proteins. It has been hypothesised that excessive sarcomeric energy consumption is an important and early factor in the pathophysiology of HCM. Therefore modulation of myocardial metabolism presents a novel target for improving myocardial performance and symptoms in patients with HCM. Trimetazidine is an anti-anginal agent which like perhexiline reduces fatty acid oxidation and increases glucose oxidation, thus increasing the efficiency of energy production. Trimetazidine has been shown to significantly improve exercise performance in patients with stable angina, ischaemic and non ischaemic cardiomyopathy, either as monotherapy or in combination with beta-blockers or calcium channel blockers,

DESIGN: A single centre prospective randomised, double blind, placebo-controlled, trial of trimetazidine therapy.

DOSING: 20 mg Trimetazidine or Placebo three times daily for three months

METHODS: The following assessments will be made at baseline and after 3 months treatment: history and physical examination, Minnesota heart failure questionnaire, fasting blood tests, electrocardiogram, echocardiogram, cardiopulmonary exercise test, six minute walk test, 24 hour ECG Holter monitor.

ELIGIBILITY:
Inclusion Criteria:

* Non-obstructive hypertrophic cardiomyopathy (gradient <30 mmHg at rest)
* NYHA (New York Heart Association) Class ≥ 2
* Peak VO2 (maximal oxygen consumption) ≤80% predicted for age and gender
* Heart rate < 90/minute at rest

Exclusion Criteria:

* Diabetes Mellitus
* Abnormal renal function (GFR<60ml/min) or hepatic impairment
* Female who is pregnant, lactating or planning pregnancy during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption | 3 months

SECONDARY OUTCOMES:
Left ventricular function | 3 months
  TDI and 2D strain
Symptom status | 3 months
  questionnaire
Arrhythmia | 3 months
  24 Hour Holter
Cardiac biomarkers | 3 months
Exercise capacity | 3 months
  6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Perry M Elliott, MBBS MD, Principal Investigator — University College, London
Locations (1):
- The Heart Hospital, UCLH, London, United Kingdom

REFERENCES:
- [Derived] Coats CJ, Pavlou M, Watkinson OT, Protonotarios A, Moss L, Hyland R, Rantell K, Pantazis AA, Tome M, McKenna WJ, Frenneaux MP, Omar R, Elliott PM. Effect of Trimetazidine Dihydrochloride Therapy on Exercise Capacity in Patients With Nonobstructive Hypertrophic Cardiomyopathy: A Randomized Clinical Trial. JAMA Cardiol. 2019 Mar 1;4(3):230-235. doi: 10.1001/jamacardio.2018.4847. PMID 30725091